CLINICAL TRIAL: NCT01608646
Title: Study of Dihydropyrimidine Dehydrogenase for Predicting Efficacy and Safety to S-1 Plus Oxaliplatin in Gastrointestinal Cancer
Brief Title: Study of DPD for Predicting Efficacy and Safety to S-1 Plus Oxaliplatin in Gastrointestinal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOTTG270105
Record Dates: First submitted 2012-05-13; First posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Gastrointestinal Cancer
Keywords: S-1; Oxaliplatin; Dihydropyrimidine Dehydrogenase
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — S 1 (combination); Oxaliplatin; titanium silicide; tegafur-gimeracil-oteracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1 plus oxaliplatin (No Intervention): S-1 40 mg/m2 administered orally BID after breakfast and evening meal from Day 1 through Day 14 with a single dose of oxaliplatin 130 mg/m2 will be administered as an 2-hour IV infusion following the morning dose of S-1 on Day 1. The combination therapy will be repeated every 3 weeks.
  Interventions: Drug: S-1 plus oxaliplatin

INTERVENTIONS:
Drug: S-1 plus oxaliplatin — S-1 40 mg/m2 administered orally BID after breakfast and evening meal from Day 1 through Day 14 with a single dose of oxaliplatin 130 mg/m2 will be administered as an 2-hour IV infusion following the morning dose of S-1 on Day 1. The combination therapy will be repeated every 3 weeks.
  Other Names: TS-1 plus oxaliplatin; Teysuno plus oxaliplatin

SUMMARY:
In this study, the relationship between DPD and the effects of S-1 combined with oxaliplatin chemotherapy were investigated in 200 patients with gastrointestinal carcinoma.

DETAILED DESCRIPTION:
A new oral DPD inhibitory fluoropyrimidine (DIF), S-1, is reportedly effective against gastrointestinal carcinoma. In this study, the relationship between activity of DPD in peripheral blood and the effects of chemotherapy were investigated in 200 patients treated with first-line S-1 combined with platinum chemotherapy for gastrointestinal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧18;
* Histologically or cytologically confirmed gastrointestinal cancer；
* ECOG ≦2;
* Physician's intention to treat with S-1 combined with platinum regimen on disease status and clinical judgment;
* Life expectancy of at least three months;
* Written informed consent to participate in the trial;

Exclusion Criteria:

* History of severe hypersensitivity reactions to the ingredients of S-1 or oxaliplatin;
* Inadequate hematopoietic function which is defined as below:

  * white blood cell (WBC) less than 3,500/mm^3
  * absolute neutrophil count (ANC) less than 1,500/mm^3
  * platelets less than 80,000/mm^3
* Inadequate hepatic or renal function which is defined as below:

  * serum bilirubin greater than 1.5 times the upper limit of normal range
  * alanine aminotransferase (ALT) or aspartate aminotransferase (AST)
  * greater than 2.5 times the ULN if no demonstrable liver metastases or
  * greater than 5 times the ULN in the presence of liver metastases
  * blood creatinine level greater than 2 times ULN
* Presence of peripheral neuropathy;
* Receiving a concomitant treatment with other fluoropyrimidine drug or flucytosine drug;
* Women who is pregnant or lactating or fertile women of child-bearing potential unless using a reliable and appropriate contraceptive method throughout the treatment period (Including male);
* Psychiatric disorder or symptom that makes participation of the patient difficult;
* Concomitant illness that might be aggregated by active, non-controlled disease such as congestive heart failure, ischemic heart disease, uncontrolled hypertension or arrhythmia with in six months;
* Severe complication(s), e.g., paresis of intestines, ileus, radiographically confirmed interstitial pneumonitis or pulmonary fibrosis, glomerulonephritis ,renal failure, poorly-controlled diabetes;
* Known DPD deficiency;
* Receiving a concomitant treatment with sorivudine or Brivudine within two months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response | Every eight weeks
  Tumor response was evaluated by RECIST 1.1. The relationship between DPD activity and the objective tumor response will be evaluated by Cox's proportional hazards regression model.

SECONDARY OUTCOMES:
Overall survival | Three year
  The relationship between DPD activity and the overall survival will be evaluated by Cox's proportional hazards regression model.
Progress-free survival | one year
  The relationship between DPD activity and the PFS will be evaluated by Cox's proportional hazards regression model.
Adverse event incidence | One year
  The relationship between DPD activity and the drug-related toxicity incidence will be evaluated by Cox's proportional hazards regression model.

CONTACTS AND LOCATIONS:
Overall Officials: WENCHAO LIU, professor, Principal Investigator — xijing hospital of the fourth military medical univercity
Locations (1):
- Xijing hospital of the fourth military medical univercity, Xijing, Shanxi, China